CLINICAL TRIAL: NCT01731418
Title: Efficacy of Narrative Exposure Therapy (NET) in a Sample of Iranian Women Exposed to Intimate Partner Violence (IPV)
Brief Title: NET in Iranian Women Suffering From Post Traumatic Stress Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tahere Orang, PhD Student, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TO-10122012-UK
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Mental Disorders; Domestic Violence
Keywords: Post Traumatic Stress Disorder; Depression; Intimate Partner violence; Narrative Exposure Therapy
MeSH Terms: conditions — Mental Disorders; Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treamtent-as-usual (Other): Treatment-as-usual can be defined as the commonly used psychotherapy for abused women in Iran, such as medical therapy and/or supportive psychotherapy.
  Interventions: Other: Treatment-as-usual
- Narrative Exposure Therapy (Experimental): Narrative Exposure Therapy (NET) is a standardized short-term approach based on the principles of cognitive behavioral exposure therapy and testimony therapy for the treatment of PTSD resulting from organized violence.
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Narrative Exposure Therapy (NET) is a treatment approach that was developed by a research group of the University of Konstanz (Schauer, Neuner, & Elbert, 2005, 2011). In NET, the patient repeatedly talks about the most arousing traumatic events in detail while re-experiencing the emotions associated with this event. In the process, the patient constructs a narration of his life, focusing on the detailed report of the traumatic experiences.
  Other Names: NET
  Arms: Narrative Exposure Therapy
Other: Treatment-as-usual — Treatment-as-usual was defined as the commonly used psychotherapy for abused women in Iran, such as medical therapy and/or supportive counseling.
  Regarding supportive counselling, the sessions included:
  Life skill education CBT techniques ACT techniques Finding resources to stop violence Discussing marital and sexual conflicts with the presence of husbands Working on their children problems Improvement of communication skills
  Arms: Treamtent-as-usual

SUMMARY:
The proposed study seeks to investigate to what extent Narrative Exposure Therapy (NET) is an effective treatment for the reduction of symptoms of Post-Traumatic Stress Disorder (PTSD) and depression and for the improvement of daily functioning in Iranian women who have experienced intimate partner violence (IPV). In addition, the study seeks to investigate whether NET therapy could lead to the reduction of Intimate Partner Violence (IPV) within their marriage.

ELIGIBILITY:
Inclusion Criteria:

* being victims of Intimate Partner Violence and seeking help at target clinics in order to reduce their psychological symptoms, currently living together with their partner/husband, meeting the set cut-off point on the PTSD scale according to DSM-IV.

Exclusion Criteria:

* schizophrenia, epilepsy, mental retardation, drug abuse and mal-nourishment

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Diagnostic Scale (PDS/PSS-I). | Symptoms will be assessed at pre-treatment-point and post-treatment-point (up to 6-month follow-ups)
  The PDS/PSS-I is a 17-item screening instrument on a 4-point-Likert-scale (0 = not at all to 3 = very much). The PDS aims at assessing all Diagnostic and Statistical Manual (DSM-IV) criteria of a Post Traumatic Stress Disorder (PTSD), and thus it includes information about the nature of the traumatic event and the level of functional interference.
The Patient Health Questionnaire-9 (PHQ-9) | At pre-treatment-point, post-treatment-point, and 3- and 6-month follow-ups
  The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module
The Hopkins Symptom Checklist-25 (HSCL-25) | At pre-treatment-point, post-treatment-point, and 3- and 6-month follow-ups
  The Hopkins Symptom Checklist 25 would be used to screen for symptoms of depression and anxiety.
Perceived Stress Scale-4 | At pre-treatment-point, post-treatment-point and 3- and 6-month follow-ups
  The Perceived Stress Scale (PSS) would be used to assess the perception of stress over the course of the last month preceding the interview

SECONDARY OUTCOMES:
Composite Abuse Scale (CAS) | At pre-treatment-point, post-treatment-point, and 3- and 6-month follow-ups
  The CAS, a 30-item validated research instrument, is a widely used self-report questionnaire of behaviors that women describe as abusive by their partners. It is a self-report measure that provides standardized sub scale scores on four dimensions of intimate partner abuse. The four dimensions are Severe Combined Abuse, Emotional Abuse, Physical Abuse, and Harassment, scaled from 0 (never) to 5 (daily) over a period of 12-month.
The Work and Social Adjustment Scale (WSAS) | At pre-treatment-point, post-treatment-point and 3- and 6-month follow-ups
  The WSAS is a widely used 5-item measure of disability. Its psychometric properties were analyzed and shown in different studies and disorders (Mataix-Cols et al, 2005; Mundt et al, 2002).
The Life Events Checklist | At pre-treatment-point, post-treatment-point and 3- and 6-month follow-ups
  The Life Events Checklist (LEC) is a brief, 17-item, self-report measure designed to screen for potentially traumatic events in a respondent's lifetime. The LEC assesses exposure to 16 events known to potentially result in PTSD or distress and includes one item assessing any other extraordinarily stressful event not captured in the first 16 items.
Checklist of family violence | At pre-treatment-point, post-treatment-point and 3- and 6-month follow-ups
  This checklist assessing the incidence of domestic violence was developed by Catani (2002) and includes questions on physical abuse, verbal violence, neglect and sexual abuse as well as witnessing intimate partner violence between parents.

OTHER OUTCOMES:
Borderline Symptom List (BSL-23) | At pre-treatment-point, post-treatment-point and 3- and 6-month follow-ups
  The BSL-23 is a shortened form of the full version of the BSL-95. The self-report questionnaire assesses borderline-specific symptomatology on a five response scale ranging from 0 (not at all) to 4 (very strongly).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, Professor, Study Chair — University of Konstanz
Locations (1):
- Mental Health Clinics, Tehran, Iran

REFERENCES:
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505